CLINICAL TRIAL: NCT06905977
Title: Long Term Follow-up Study on Thick Cornea with High Back Elevation
Brief Title: Thick Cornea with High Back Elevation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Magdy Fily, Principle investigator, Assiut University
Other Study IDs: Thick cornea
Record Dates: First submitted 2025-03-14; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Corneal Thickness Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: pentacam — we will follow up on cases of thick cornea with high back elevation

SUMMARY:
To follow up cases of thick cornea with high back elevation by pentacam.

DETAILED DESCRIPTION:
The cornea plays a crucial role in refraction and so help in good visual acuity. with its thickness and back elevation being essential parameters in diagnosing and managing corneal diseases such as keratoconus.

The normal human cornea has a central thickness of approximately 540-550 µm. The periphery is generally thicker, reaching up to 700 µm. Corneal thickness is influenced by genetics, hydration, and intraocular pressure.Thick Cornea (> 540 µm): Seen in conditions such as corneal edema and Fuchs' dystrophy. Thin Cornea (< 500 µm): Observed in keratoconus, LASIK-induced thinning, and corneal ectasia.

Back corneal elevation is assessed using corneal topography or tomography, typically referenced to a best-fit sphere (BFS). In normal cases, Back corneal elevation is usually ≤12 µm above the BFS, indicating a structurally healthy cornea without signs of ectasia. Susceptible elevation ranges between 12-20 µm, which may be an early indicator of corneal instability, such as subclinical keratoconus. Therefore, it should be evaluated alongside other parameters, including pachymetry, anterior curvature, and biomechanical properties. Abnormal back corneal elevation is generally considered >20 µm, particularly if localized or asymmetric, and is strongly associated with corneal ectatic disorders such as keratoconus, pellucid marginal degeneration, or post-LASIK ectasia. This abnormal elevation is often accompanied by other risk factors, including increased posterior corneal curvature, corneal thinning, and significant asymmetry, necessitating further assessment and monitoring.

Many cases of thick cornea are associated with high back elevation and this discourage refractive surgery in such cases so in investigator's study the investigator will follow up these cases to determine if these corneas are considered normal corneas or not.

ELIGIBILITY:
Inclusion Criteria:

Any patient can interact with pentacam. Both Genders: include both males and females. Patients with thick cornea (>540 µm) with high back elevation.

Exclusion Criteria:

* Patients with any eye disease (significant cataract or unstable glaucoma)
* Uncontrolled external disease such as blepharitis , moderate to severe dry eye and allergy.
* Patient with ocular disease such as uveitis, post herpetic infection and corneal opacity

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: any age can interact with pentacam device
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of corneal thickness and back corneal elevation by pentacam device | Baseline
  The investigator will image the cornea to measure corneal thickness and back corneal elevation using the Pentacam device and follow up for cases of thick corneas with high back elevation at 3 months, 6 months, and 1 year.